CLINICAL TRIAL: NCT04582461
Title: Role of Preoperative Multislice Computed Tomography to Predict the Risk of Pancreatic Fistula After Whipple's Operation.
Brief Title: Role of Preoperative Multislice Computed Tomography in Whipple's Operation.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelbaset Mahmoud Mohamed, Principal investigator, Assiut University
Other Study IDs: multislice computed tomography
Record Dates: First submitted 2020-09-23; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula | interventions — Multidetector Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: multislice computed tomography — All patients will undergo a preoperative multiphasic multidetector CT scan before surgery.The unenhanced scan will be used to generate a CT reconstruction of the upper abdomen (from the diaphragm to the kidneys) with a 5mm thickness. Two different radiologists (D.F. and D.I.), blinded to patient information, measured total fat volume (TFV), visceral fat volume (VFV), and analyzed pixels with densities in the - 190 hounsfield units (HU) to - 20 HU range. the ratio between the density of the pancreas over the density of the spleen will be calculated and the maximum diameter of the pancreatic duct will be measured using the arterial phase in order to better identify the entire length of the duct.

SUMMARY:
Preoperative assessment of visceral fat volume(VFV),total fat volume(TFV),pancreas/spleen density ratio and pancreatic duct diameter by multislice computed tomography abdomen to predict the risk of pancreatic fistula after Whipple's operation.

DETAILED DESCRIPTION:
pancreatic cancer has ranked the 11th most common cancer in the world and seventh leading cause of cancer-related deaths worldwide. Worldwide incidence and mortality of pancreatic cancer correlate with increasing age and is slightly more common in men than in women(1).

There are many risk factors for pancreatic cancer, such as age, tobacco smoking, heavy alcohol consumption, obesity, low physical activity, chronic pancreatitis, long-standing type 2 diabetes, ABO blood type, and family history(2).

Pancreatic cancer is mainly divided into two types of pancreatic cancer: pancreatic adenocarcinoma, which is the most common (85% of cases) arising in exocrine glands of the pancreas, and pancreatic neuroendocrine tumor (PanNET), which is less common (less than 5%) and occurs in the endocrine tissue of the pancreas.Signs and symptoms of pancreatic cancer often don't occur until the disease is advanced(3).

Upon progression of the tumor, it manifests as a gradual onset of non-specific symptoms including jaundice, weight loss, light-colored stools, abdominal pain and fatigue(4).

Treatment for pancreatic cancer depends on the stage and location of the cancer as well as on your overall health and personal preferences. Surgery, chemotherapy and radiotherapy are traditionally used to extend survival and/or relieve the patients' symptoms. However, for advanced-stage cancer cases, there is still no definite cure(5).

Postoperative pancreatic fistula (POPF) remains one of the most frequent and threatening complication after pancreatoduodenectomy (PD). The occurrence ranges from 10% to 30%(6).

Depending on its severity, it may be responsible for distant organ dysfunction and subsequent mortality, prolonged length of in-hospital stay, and increased health care costs(7).

Both prevention and treatment of POPF are challenging. Among the potential strategies to reduce the incidence and the severity of POPF, different surgical techniques(8) have been proposed along with the perioperative inhibition of exocrine pancreatic secretion(9).

An additional key factor to improve patient management may be to find reliable means of calculating and predicting the risk of POPF. The ability of anticipating the risk of POPF before surgery based on peculiar patient features might establish a more customized preoperative program for patients with high risk of fistula, potentially excluding subjects with elevated risk from surgical resection or to set up protocols for a strict and early detection of warning clinical scenario .Previous studies and reviews described different variables correlated to the occurrence of POPF, in particular, patient characteristics such as American Society of Anesthesiology score, body mass index, age, malnutrition, muscle cachexia, medical history and morbidities(10)(11)and intraoperative findings, that is, small Wirsung duct diameter, soft pancreatic texture, and estimated blood loss(12).

The multivariate analysis revealed that a visceral fat volume(VFV) >2334 cm3,total fat volume(TFV) >4408 cm3, pancreas/spleen density ratio <0.707, and pancreatic duct diameter <5mm were predictive of POPF(13).

Also baseline radiological findings, such as fat distribution, radiological characteristics of abdominal skeletal muscles, estimated pancreatic remnant volume, and pathway of the enhancement attenuation have been correlated with the risk of complication development and POPF, but with inconsistent results(14)(15).

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to the radiology department for multislice computed tomography Abdomen examination for preoperative evaluation before Whipple's operation over the estimated period of the study.

Exclusion Criteria:

* Patients with contraindications to multislice computed tomography as a history of reactions to contrast agents, radioactive iodine treatment for thyroid disease, metformin use, and chronic or acutely worsening renal disease.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Selection of average 100 patients expected to visit Assiut university hospitals for multislice computed tomography Abdomen before Whipple's operation according to the recorded flow on the Picture Archiving and Communication System (PACS) in the last year.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
preoperative prediction of occurence of pancreatic fistula after Whipple's operation to enhance surveillance and further management as early as possible. | Baseline
  Preoperative assessment mainly abdominal fat distribution (expressed in centimeter cubic) by multislice computed tomography abdomen to predict the risk of pancreatic fistula after Whipple's operation.

REFERENCES:
- [Background] Ilic M, Ilic I. Epidemiology of pancreatic cancer. World J Gastroenterol. 2016 Nov 28;22(44):9694-9705. doi: 10.3748/wjg.v22.i44.9694. PMID 27956793
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Hidalgo M, Cascinu S, Kleeff J, Labianca R, Lohr JM, Neoptolemos J, Real FX, Van Laethem JL, Heinemann V. Addressing the challenges of pancreatic cancer: future directions for improving outcomes. Pancreatology. 2015 Jan-Feb;15(1):8-18. doi: 10.1016/j.pan.2014.10.001. Epub 2014 Oct 17. PMID 25547205
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Mohammed S, Van Buren G 2nd, Fisher WE. Pancreatic cancer: advances in treatment. World J Gastroenterol. 2014 Jul 28;20(28):9354-60. doi: 10.3748/wjg.v20.i28.9354. PMID 25071330
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Enestvedt CK, Diggs BS, Cassera MA, Hammill C, Hansen PD, Wolf RF. Complications nearly double the cost of care after pancreaticoduodenectomy. Am J Surg. 2012 Sep;204(3):332-8. doi: 10.1016/j.amjsurg.2011.10.019. Epub 2012 Mar 29. PMID 22464011
- [Background] Huttner FJ, Fitzmaurice C, Schwarzer G, Seiler CM, Antes G, Buchler MW, Diener MK. Pylorus-preserving pancreaticoduodenectomy (pp Whipple) versus pancreaticoduodenectomy (classic Whipple) for surgical treatment of periampullary and pancreatic carcinoma. Cochrane Database Syst Rev. 2016 Feb 16;2(2):CD006053. doi: 10.1002/14651858.CD006053.pub6. PMID 26905229
- [Background] Koti RS, Gurusamy KS, Fusai G, Davidson BR. Meta-analysis of randomized controlled trials on the effectiveness of somatostatin analogues for pancreatic surgery: a Cochrane review. HPB (Oxford). 2010 Apr;12(3):155-65. doi: 10.1111/j.1477-2574.2010.00157.x. PMID 20590882
- [Background] Lermite E, Pessaux P, Brehant O, Teyssedou C, Pelletier I, Etienne S, Arnaud JP. Risk factors of pancreatic fistula and delayed gastric emptying after pancreaticoduodenectomy with pancreaticogastrostomy. J Am Coll Surg. 2007 Apr;204(4):588-96. doi: 10.1016/j.jamcollsurg.2007.01.018. Epub 2007 Mar 2. PMID 17382217
- [Background] Lin JW, Cameron JL, Yeo CJ, Riall TS, Lillemoe KD. Risk factors and outcomes in postpancreaticoduodenectomy pancreaticocutaneous fistula. J Gastrointest Surg. 2004 Dec;8(8):951-9. doi: 10.1016/j.gassur.2004.09.044. PMID 15585382
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Sandini M, Bernasconi DP, Ippolito D, Nespoli L, Baini M, Barbaro S, Fior D, Gianotti L. Preoperative Computed Tomography to Predict and Stratify the Risk of Severe Pancreatic Fistula After Pancreatoduodenectomy. Medicine (Baltimore). 2015 Aug;94(31):e1152. doi: 10.1097/MD.0000000000001152. PMID 26252274
- [Background] Kirihara Y, Takahashi N, Hashimoto Y, Sclabas GM, Khan S, Moriya T, Sakagami J, Huebner M, Sarr MG, Farnell MB. Prediction of pancreatic anastomotic failure after pancreatoduodenectomy: the use of preoperative, quantitative computed tomography to measure remnant pancreatic volume and body composition. Ann Surg. 2013 Mar;257(3):512-9. doi: 10.1097/SLA.0b013e31827827d0. PMID 23241871
- [Background] McAuliffe JC, Parks K, Kumar P, McNeal SF, Morgan DE, Christein JD. Computed tomography attenuation and patient characteristics as predictors of complications after pancreaticoduodenectomy. HPB (Oxford). 2013 Sep;15(9):709-15. doi: 10.1111/hpb.12037. Epub 2013 Jan 10. PMID 23458275